CLINICAL TRIAL: NCT02765659
Title: A Community-based Implementation Model for HIV Prevention and Testing in Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Kamuzu College of Nursing, University of Malawi (Unknown); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Kathy Norr, Professor Emerita, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-0691; R01NR015409 (NIH)
Record Dates: First submitted 2016-04-23; First posted 2016-05-06 (Estimated); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: HIV CDC Category A1
Keywords: HIV; Prevention; Implementation; Community based participatory research

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Community 1 (Other): Receives Mzake ndi Mzake T1 immediately after baseline
  Interventions: Behavioral: Mzake ndi Mzake T1
- Community 2 (Other): Receives Mzake ndi Mzake T2 immediately after Post-T1 evaluation
  Interventions: Behavioral: Mzake ndi Mzake T2
- Community 3 (Other): Receives Mzake ndi Mzake T3 immediately after Post-T2 Evaluation
  Interventions: Behavioral: Mzake ndi Mzake T3

INTERVENTIONS:
Behavioral: Mzake ndi Mzake T1 — a 6-session peer group intervention focusing on primary HIV prevention and early testing and entry to treatment for secondary prevention - offered immediately after baseline
  Arms: Community 1
Behavioral: Mzake ndi Mzake T2 — a 6-session peer group intervention focusing on primary HIV prevention and early testing and entry to treatment for secondary prevention - offered immediately after post-T2 evaluation
  Arms: Community 2
Behavioral: Mzake ndi Mzake T3 — a 6-session peer group intervention focusing on primary HIV prevention and early testing and entry to treatment for secondary prevention - offered immediately after post-T3 evaluation
  Arms: Community 3

SUMMARY:
This implementation study is testing whether community members can use a 3-step model (prepare, roll-out and sustain) to implement an efficacious peer group HIV prevention intervention with fidelity and effectiveness in a single district in Southern Malawi. A collaborative partnership including university researchers and district government, health system and traditional leaders will support community volunteers in implementation. Both the implementation process and the effectiveness of the intervention when implemented by communities will be evaluated.

DETAILED DESCRIPTION:
In response to the National Institutes of Health's call for empirically-supported models to implement research-tested health behavior change interventions, the investigators are testing a 3-step (prepare, roll-out, and sustain) Community Implementation Model (Model) in low-resource African communities. The Model is adapted from a theory-based model that was effective in implementing a hospital-based intervention in South Africa. Its participatory approach, clear steps, observable benchmarks and multimedia Toolkit will facilitate community ownership and build capacity to use the Model with fidelity. The investigators test whether community members can use the Model to effectively implement a peer group HIV prevention intervention called Mzake ndi Mzake (Friend to Friend) with fidelity and effectiveness. Developed and tested among several populations in Malawi (R01-NR08058), This intervention was efficacious in rural, central Malawi. Intervention communities had significantly better outcomes, including higher condom use and HIV testing for both adults and adolescents, than control communities. The investigators evaluate the Model's implementation success in Phalombe District, in southern Malawi, where the HIV prevalence of 14.5% is twice that of other regions. Our implementation partnership builds on the strengths and contributions of four sectors. Traditional community leaders mobilize their communities' assets, including volunteers to implement the peer group intervention. The District health system has formal authority in health organizations, contributes health knowledge, and provides local District health data. The District political administration supports this effort by negotiating donated space for an HIV/AIDS Resource Centre and by pledging funds to sustain and expand implementation of the intervention if communities demonstrate that they can use the Model. Researchers from both US and Malawi universities contribute the Model and the Mzake ndi Mzake peer group intervention, provide supportive technical assistance for program implementation and conduct evaluations. Specific aims and their evaluation are: Aim 1) Prepare and support 3 communities in using the Model to implement Mzake, evaluated with community self-rated benchmarks. Aim 2) Identify implementation patterns across sites and over time, evaluated using mixed-methods to integrate benchmarks with observations, focus groups, and interview. Aim 3) Assess communities' effectiveness in using the Model to implement Mzake, evaluated with a stepped wedge design (N = 864). Analysis uses multi-level hierarchical models to detect improvements over time in HIV-related behavioral outcomes and a symptoms interview with a nurse for sexually transmitted infections (STIs) in participants who have received the intervention compared to the delayed-intervention control group. (Our original plan to use rapid STI tests appropriate for community use had to be modified because of new data indicating unacceptable reliability and withdrawal of one test from the market). Aim 4) Evaluate whether the Model is feasible, acceptable, effective and sustainable when used by communities to implement Mzake, examined by integrating data from Aims 1-3. If successful, this study will advance implementation science by providing a replicable evidence-based model for implementation of HIV prevention interventions and other health interventions by low-resource communities.

ELIGIBILITY:
Inclusion Criteria:

* reside in specified community,
* parental permission if under age 18

Exclusion Criteria:

* not in designated community

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1353 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Reported condom use in the last 2 months | Change from baseline up to 33 months to 33 months
  If used condoms (always, sometimes, never) in last 2 months with all sexual partners

SECONDARY OUTCOMES:
HIV test in last 12 months | Change from baseline up to 33 months
  up to 33 months If reports having an HIV test in the last 12 months
Reported sexually transmitted infection (STI) symptoms | Change from baseline up to 33 months
  STI symptoms reported during the last week in an interview with a nurse
Reported high-risk behaviors in the last 2 months | Change from baseline up to 33 months
  Number of risky behaviors: unprotected sex, sex for money, sex while drinking, multiple partners, STI symptoms or positive test
condom used at last intercourse | Change from baseline up to 33 months
  if reported using a condom the last time had sexual intercourse

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen F. Norr, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Phalombe district communitie, Phalombe, Malawi

IPD SHARING:
Plan to Share IPD: No
De-identified data will be made available to other researchers for secondary analyses after the primary outcome publications have been accepted for publication, approximately 3 years after the grant ends.

REFERENCES:
- [Background] Jere DLN, Banda CK, Kumbani LC, Liu L, McCreary LL, Park CG, Patil CL, Norr KF. A hybrid design testing a 3-step implementation model for community scale-up of an HIV prevention intervention in rural Malawi: study protocol. BMC Public Health. 2018 Aug 2;18(1):950. doi: 10.1186/s12889-018-5800-3. PMID 30071866
- [Derived] Norr KF, Banda CK, Chang C, Krishna S, Kumbani LC, Liu L, McCreary LL, Patil CL. Condom use increased after a peer group intervention implemented by community volunteers in Malawi. BMC Public Health. 2024 Jun 3;24(1):1483. doi: 10.1186/s12889-024-18991-z. PMID 38831266
- [Derived] Norr KF, Banda CK, Chang C, Krishna S, Kumbani LC, Liu L, McCreary LL, Patil CL. Condom use increased after a peer group intervention implemented by community volunteers in Malawi. Res Sq [Preprint]. 2023 Jul 4:rs.3.rs-3120974. doi: 10.21203/rs.3.rs-3120974/v1. PMID 37461672
- [Derived] Kumbani LC, Jere DL, Banda CK, Chang C, Liu L, McCreary LL, Patil CL, Norr KF. A peer group intervention implemented by community volunteers increased HIV prevention knowledge. BMC Public Health. 2023 Feb 10;23(1):301. doi: 10.1186/s12889-022-14715-3. PMID 36765344